CLINICAL TRIAL: NCT01027091
Title: The Study of a Safe and Cost-effective Method to Identify Patients at Low Risk for the Development of Significant Hypocalcemia After Total Thyroidectomy.
Brief Title: The Study of a Safe and Cost-effective Method to Identify Patients at Low Risk of Significant Hypocalcemia After Total Thyroidectomy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G. Hatzikosta General Hospital (Other)
Responsible Party: George A. Economou resident of G.Hatzikosta G.H Surgery Department, G.Hatzikosta General Hospital
Other Study IDs: 7/06-11-09
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-11

CONDITIONS: Hypocalcemia After Total Thyroidectomy
Keywords: hypocalcemia; total thyroidectomy
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients with positive slope: patients with positive slope in the levels of free serum calcium levels between 6th and 12th postoperative hour
- patients with negative or no slope: patients with negative or no slope in the levels of free serum calcium levels between 6th and 12th postoperative hour.

SUMMARY:
Hypocalcemia is the complication, after total thyroidectomy, that usually determines the length of hospital stay.Serum calcium levels is a quick and cost-effective practice to recognise hypocalcemia in the postoperative follow up.

OBJECTIVE: The objective of this perspective study is to determine if consecutive postoperative serum calcium levels early after total thyroidectomy can be used to identify patients who are unlikely to develop significant hypocalcemia and can be safely discharged within 24 to 48 hours postoperative.

DETAILED DESCRIPTION:
INTRODUCTION:

In recent years there has been a global trend towards more radical and aggressive approach to thyroid surgery (total or subtotal thyroidectomy against semithyreoeidectomy), almost regardless of the pathological cause, even for benign diseases. There is also developed, a serious skepticism as complications of total or subtotal thyroidectomy is neither rare nor insignificant. In particular, complications of thyroidectomy is the laryngeal nerve paresis (0.2% bilateral, unilateral 3,7-3,9%, 2% transient, lasting 1%), bleeding (1-2%), infection of the wound (0, 3-1,6%) and hypocalcaemia (permanent hypocalcaemia in over 6 months follow up 1,7-4,4%, while transient, manageable with vit D and calcium substitution 8,3-9,9%). The post total thyroidectomy hypocalcaemia is not only more frequent but also has the most delayed onset after surgery (up to several 24hours later) in relation to bleeding and paresis of the laryngeal nerve, which is immediate postoperative complications. This is the main cause of prolonged hospitalization and monitoring of patients postoperatively which is linked to increased risk of bacterial infections and increased cost.9, 10 Great effort has been made in the last 15 years to reduce the length hospital stay of patients in order to perform the total thyroidectomy as a one day surgery.6, 11 In this way great importance is the prediction of those patients are more likely to experience post-operative hypocalcaemia. The appearance of postoperative hypocalcaemia associated with specific diseases such as thyroid disease Graves, the thyreotoxicosis and thyroid cancer 7.8, and the surgical technique (the extent of excision, the type of thyroid artery ligation, the number of parathyroid recognized intraoperative but also those autotransplanted) 12. Moreover, beyond these factors, great importance is given to methods of monitoring patients to find reliable indicators to allow safe release out of the hospital after the first 24 hours without risk of hypocalcaemia. The measurement of parathyroid hormone (PTH) both intraoperative and postoperatively (4 hours) is a hot topic in contemporary literature and promises accurate predictions 13, but there is disagreement about the precise time of receiving the specimens and great consideration about the increased cost 14, 15 (at our hospital is not even available). An older, simple, fast and economical method is to measure levels of free serum calcium 6,9. Despite that the correlation of the immediate post-operative levels of free calcium, with the likelihood of developing hypocalcaemia has variations in different surveys, resulting to early release of patients directly when free calcium is in normal range, by some departments, while others follow strict protocols of monitoring patients for days . However, the variation in the levels of free serum calcium between the first 6 and 12 postoperative hours alone or in combination with measurement of PTH seems to give some answers and it is under great consideration in the international community.

It is therefore, in line with the current literature, important to develop a safe, and also cost-effective protocol monitoring patients after total thyroidectomy, which, in combination with predisposing risk factors of hypocalcaemia, will predict low-risk patients for developing hypocalcaemia and allow secure release from the hospital.

PRIMARY OBJECTIVES:

The objective of this perspective study is to correlate the variability of the levels of free serum calcium (Ca + +), and also the levels of albumin (ALB), phosphorus (PO-3), magnesium (Mg) and total albumin (TPR), between two measurements on 6 and 12 hours postoperatively, the incidence of hypocalcaemia in patients undergoing total thyroidectomy for any reason. The aim is to develop on the basis of variation in levels of free serum calcium, a secure method of prediction and identification of low risk patients for developing hypocalcaemia providing an early release from hospital.

SECONDARY OBJECTIVES:

The correlation between development of hypocalcaemia in patients after total thyroidectomy with the following factors:

* Gender,
* Age,

Intraoperative factors:

* Intraoperative recognition of parathyroid glands
* Possible autotransplantation of parathyroid glands
* Using scissors, ultrasonic Ligasure compared using ultrasonic scissors
* use Ultracision ligation
* Use of hemostatic
* Volume of blood loss;
* Volume and weight; preparation

Postoperative factors based on the histological-pathological report:

-Underlying thyroid pathology

CHOICE / NUMBER OF PATIENTS:

At least 80 patients with any thyroid pathology undergoing a total thyroidectomy regardless of gender, age and medication preceding the one exception, patients treated with substitutes calcium and vitamin D.

METHODS (CLINICAL-LABORATORY) The hypocalcaemia is defined in the study as clinical hypocalcaemia. Required symptoms of hypocalcaemia are regional or perioral numbness and signs of hypocalcaemia: Trousseau sign (karpopodic spasm) and Chvostek sign (spasm CN VII) and / or the levels of free serum calcium below 0,5 mg / dl lower than the normal price laboratory (8,2-10,6 mg / dl).

Each patient included in the study is provided with:

* Detailed preoperative history and physical examination. Recording; all preoperative examinations before the introduction of the clinical (U / S thyroid scan, FNA biopsy)
* Receiving laboratory examinations

  * Preoperative
  * on the 6th, 12th and 24th postoperative hours,
  * every 24 hours after the first 24 hours as long a patient remains in clinical
  * at least 7 days after hospital discharge
* The laboratory control, includes

  1. pre-operatively and 6hr postoperatively :

     * Complete blood count,
     * levels of urea,
     * creatinine,
     * sodium potassium,
     * glucose, -
     * albumin,
     * total protein, -
     * transaminases,
     * γ-GT,
     * total and immediate cholerethrini,
     * alkaline phosphatase,
     * lactate dehydrogenase,
     * amylase,
     * free serum calcium,
     * phosphorus,
     * magnesium
  2. Ιn all other measurements:

     * Free serum calcium,
     * phosphorus,
     * magnesium,
     * albumin and
     * total albumin levels
* Surgery information, detailed references of:

  1. The time of onset and completion of surgery
  2. The use of ligation, Ligasure ultrasonic scissors or Harmonic
  3. The recognition of intraoperative parathyroid glands, their number and their potential autologous transplants
  4. The weight of the specimen
  5. The blood loss (large or small)
  6. The use of hemostatics
  7. The use neuromonitoring
  8. The type of antibiotics used
  9. The technical rehabilitation of the skin and the use of skin glue
  10. The installation of vacuum drainage
* Detailed list of all medication received by the patient during hospitalization
* No intravenous or oral calcium or vitamin D supplementation before completing 12 hours postoperatively except the clinical case of development of significant hypocalcaemia.
* Detailed clinical examination, including:

  1. Testing for Regional numbness
  2. Monitored for signs of Chvostek and Trousseau
  3. Detailed analysis of the histological-pathological report with a detailed record of findings of the final pathology of the thyroid.

ELIGIBILITY:
Inclusion Criteria:

* patients with any thyroid pathology undergoing total thyroidectomy regardless of gender, age and medication

Exclusion Criteria:

* patients treated with substitutes calcium and vitamin D.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with any thyroid pathology undergoing total thyroidectomy regardless of gender, age and medication
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-06 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of the variability of the levels of free serum calcium (Ca + +), between two measurements on 6 and 12 hours postoperatively, the incidence of hypocalcaemia in patients undergoing total thyroidectomy for any reason. | 6hr, 12hr, 24hr, 48hr postopreratively

SECONDARY OUTCOMES:
The correlation between development of hypocalcaemia in patients after total thyroidectomy with the following factors: · Gender, · Age,
The correlation between development of hypocalcaemia and the Intraoperative recognition of parathyroid glands and possible autotransplantation of parathyroid glands,
The correlation between development of hypocalcaemia in patients after total thyroidectomy with the Underlying thyroid pathology based on the histological-pathological report:
The correlation between development of hypocalcaemia in patients after total thyroidectomy with the following factors: Use of Ligasure use of Ultracision, Use of hemostatic,Volume of blood loss, Volume and weight of specimen

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos K Tsimoyiannis, DR, MD, FACS, FABI,, Study Director — G. Hatzikosta General Hospital
Locations (1):
- G.Hatzikosta General Hospital, Ioannina, Ioannina, Greece